CLINICAL TRIAL: NCT05783908
Title: Impact of Non-magnetic Screen Respiratory Self-guidance During MRI-guided Radiotherapy Sessions for Mobile Lesions
Acronym: RespEcran
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022-A02774-39
Record Dates: First submitted 2023-02-10; First posted 2023-03-24 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Patient With Radiotherapy (Linac MRI); Mobile Cancerous Lesion
Keywords: Linac IRM; Pancreatic cancer; Liver cancer; Kidney cancer; Adrenal cancer; Lung cancer; Adenopathy above or below the diaphragm
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Kidney Neoplasms; Adrenal Gland Neoplasms; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without Non-magnetic screen (No Intervention): Radiotherapy treatment with Linac MRI without non-magnetic shielding
- With non-magnetic screen (Experimental): Radiotherapy treatment with Linac MRI with non-magnetic screen
  Interventions: Combination Product: With non-magnetic screen

INTERVENTIONS:
Combination Product: With non-magnetic screen — Radiotherapy treatment with Linac MRI is performed with a non-magnetic screen that will guide the patient to block the breathing
  Arms: With non-magnetic screen

SUMMARY:
The patients eligible for the study are those treated by radiotherapy on Linac MRI for a mobile cancerous lesion (pancreas, liver, kidneys, adrenals, lung, adenopathy above or below the diaphragm ...).

After signing the consent form, each patient will be randomized to one of two treatment arms:

* Standard arm : Radiotherapy treatment with Linac MRI without non-magnetic shielding
* Experimental arm : radiotherapy treatment with Linac MRI with non-magnetic screen The aim is to evaluate the effect of using a non-magnetic screen visible to the patient in the bunker during radiotherapy sessions delivered by Linac MRI on decreasing the ratio between the actual treatment time and the treatment time predicted by the machine.

DETAILED DESCRIPTION:
The patients eligible for the study are those treated by radiotherapy on Linac MRI for a mobile cancerous lesion (pancreas, liver, kidneys, adrenals, lung, adenopathy above or below the diaphragm ...).

After signing the consent form, each patient will be randomized to one of two treatment arms:

* Standard arm : Radiotherapy treatment with Linac MRI without non-magnetic shielding
* Experimental arm : radiotherapy treatment with Linac MRI with non-magnetic screen

The aim is to compare the effect of the non-magnetic screen on the blocking of the patient's breathing versus the current procedure (the blocking of the breathing is informed by the staff)

The patients will each receive 5 sessions of radiotherapy on Linac MRI. 100 patients are expected to participate in this study

Before each session will be assessed for anxiety and stress. After each session will be evaluated patient satisfaction, pain intensity and respiratory effort.

The duration of the treatment and therefore of the follow-up of the patient in the study is 1 to 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patient starting radiotherapy on Linac MRI for a mobile cancerous lesion most often in the pancreas, liver, kidneys, adrenals, lung, supra or subdiaphragmatic adenopathy
* Patient affiliated to the social security system

Exclusion Criteria:

* Patient with lesions not detected by the device's tracking system
* Patient with visual disturbances
* Contraindications to treatment with Linac MRI (epileptic patients, pregnant or breastfeeding women, metallic prosthesis or pacemaker not compatible with MRI)
* Patients with cognitive disorders
* Persons deprived of liberty or under guardianship (including curatorship)
* Pregnant or nursing woman
* Refusal to participate in the study

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-09-27 (Estimated); Study Completion 2025-09-27 (Estimated)

PRIMARY OUTCOMES:
The effect of the non-magnetic screen during radiotherapy (Change in ratio of actual treatment time to the treatment time predicted by the machine). | During 25 months
  To evaluate the effect of a non-magnetic screen visible to the patient in the bunker during radiation therapy sessions delivered by Linac MRI on decreasing the ratio of actual treatment time to the treatment time predicted by the machine.

SECONDARY OUTCOMES:
Patient respiratory effort with visual analog scale | During 25 months
  Patient respiratory effort for each radiotherapy session according to randomization arm.
  The scale is graduated from 0 to 10 with 10 = maximum respiratory discomfort and 0 = no respiratory discomfort
The positional pain with visual analog scale | During 25 months
  Compare the positional pain associated with setting up on the treatment table for each radiation therapy session according to the randomization arm.
  The scale is graduated from 0 to 10 with 0 = absence of pain and 10 = maximum pain
Level of anxiety/stress evaluated with the Spielberg scale via the STAI-Y-form grid | During 25 months
  To assess the average level of anxiety/stress for each radiation therapy session according to the randomization arm. The Spielberg scale via the STAI-form Y-A grid is used before each treatment session in order to follow the evolution of the patients' emotional state.
  20 questions with 4 possible answers : 1/ Not at all, 2/ A little, 3/Moderately , 4/ A lot.
The potential time | During 25 months
  Evaluate whether the potential time savings in screen time compensates for the time spent learning the screen during the simulation.
The patient satisfaction evaluated with an ad-hoc questionnaire. | During 25 months
  The patient's satisfaction with his or her involvement in the treatment process will be evaluated at the end of the 5 radiotherapy sessions using an ad-hoc questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges-François Leclerc, Dijon, Côte d'Or, France